CLINICAL TRIAL: NCT02415790
Title: A 4-Part, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics of E2027 in Healthy Adult, Elderly and Japanese Subjects, and the Pharmacodynamics in Healthy Adult Subjects
Brief Title: Study to Assess the Safety, Tolerability, Pharmacokinetics of E2027 in Healthy Adult and Elderly Subjects, and the Pharmacodynamics in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2027-A001-001
Record Dates: First submitted 2015-03-11; First posted 2015-04-14 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Healthy Participants
Keywords: E2027; Healthy Adult and Elderly Subjects; Pharmacokinetics/Pharmacodynamics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part A: PK of E2027 in healthy adults (Experimental): Part A consists of 6 sequential cohorts of healthy adults. There will be 8 participants in each cohort, with 6 participants randomized to E2027 and 2 participants to placebo.
  Interventions: Drug: E2027; Drug: E2027 matching placebo
- Part B: PK and PD of E2027 in healthy adults (Experimental): Part B consists of 4 sequential cohorts of healthy adult participants. There will be 8 participants in the 1st cohort, with 6 participants randomized to E2027 and 2 participants to placebo. In the 2nd to 4th cohorts, there will be 7 participants in each cohort, with 6 participants randomized to E2027 and 1 participant to placebo. Participants in the 2nd cohort will then receive placebo/the same dose of E2027 again after their washout period in the fed state for the evaluation of food effect.
  Interventions: Drug: E2027; Drug: E2027 matching placebo
- Part C: PK of E2027 in elderly cohorts (Experimental): In Part C, 1 cohort of 8 healthy elderly participants will be enrolled, with 6 participants randomized to E2027 and 2 participants to placebo.
  Interventions: Drug: E2027; Drug: E2027 matching placebo
- Part D: PK of E2027 in healthy Japanese adults (Experimental): In Part D, there will be 3 cohorts of 7 healthy adult Japanese participants, with 6 participants randomized to E2027 and 1 participant to placebo.
  Interventions: Drug: E2027; Drug: E2027 matching placebo

INTERVENTIONS:
Drug: E2027 — Part A: E2027 capsules will be administered orally in doses of 10 mg to 1200 mg in Part A and in Part B, C, and D at doses not exceeding the highest dose achieved in Part A.
Drug: E2027 matching placebo — E2027 matching placebo capsule will be administered.

SUMMARY:
This first-in-human study, designed to assess the safety, tolerability, and pharmacokinetics (PK) of single oral ascending doses of E2027, will be administered to healthy adult participants to determine the maximum tolerated dose (MTD). Thereafter, the pharmacodynamic (PD) effects of single doses of E2027 on elevation of cerebrospinal fluid (CSF) cyclic guanidine monophosphate (cGMP) in healthy adult participants will be evaluated across a broad dose range, to establish the PK/PD relationship.

DETAILED DESCRIPTION:
The study will consist of 4 parts, Parts A, B, C, and D. Part A is a single ascending dose (SAD) clinical pharmacology for evaluation of safety, tolerability, and PK characteristics up to the MTD in healthy adult (greater than or equal to 18 years and less than or equal to 50 years old). In Part B, the PK and PD effects of E2027 on CSF cGMP are evaluated in healthy adult (greater than or equal to 18 years and less than or equal to 50 years old). Participants in 2nd cohort of Part B will participate in the evaluation of food effect in Treatment Period 2. In Part C, the design is similar to Part A. This healthy elderly cohort (greater than or equal to 65 years and less than or equal to 85 years old) will provide bridging PK, safety, and tolerability data on E2027 compared to younger healthy participants in Part A and Part B. Part D will be conducted in healthy Japanese adult participants (greater than or equal to 20 years and less than or equal to 50 years old) and is designed to bridge the PK, safety, and tolerability data of E2027 between Japanese and non-Japanese participants. All parts of the study will have 2 phases: the Prerandomization Phase and the Randomization Phase. The Prerandomization Phase will consist of a Screening Period and a Baseline Period during which each participant's study eligibility will be determined and baseline assessments will be conducted. The Randomization Phase will consist of the Treatment Period and a Follow-Up Period. During the Treatment Period, participants will be randomized to receive a single oral dose of either E2027 or placebo matching E2027.

ELIGIBILITY:
Inclusion Criteria:

Part A and B only:

1. Nonsmoking, male or female, age greater than or equal to 18 years and less than or equal to 50 years old at the time of informed consent

   Part C only:
2. Nonsmoking, male or female, age greater than or equal to 65 years and less than or equal to 85 years old at the time of informed consent

   Part D only:
3. Nonsmoking, male or female, age greater than or equal to 20 years and less than or equal to 50 years old at the time of informed consent
4. Born in Japan to Japanese parents and grandparents of Japanese descent
5. Been living outside Japan for less than 5 years
6. Lifestyle, including diet, has not changed significantly since leaving Japan

   All parts:
7. Body mass index (BMI) greater than or equal to 18 and less than or equal to 30 kg/m2 at Screening

Exclusion Criteria:

1. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing
2. Females who are breastfeeding or pregnant at Screening or Baseline
3. If females of childbearing potential who:

   1. Had unprotected sexual intercourse within 30 days before study entry and do not agree to use a highly effective method of contraception
   2. Are currently abstinent, and do not agree to use a double barrier method or refrain from sexual activity
4. Males who have not had a successful vasectomy (confirmed azoospermia) or they and their female partners do not meet the criteria above. No sperm donation is allowed during the study period or for 28 days after study drug discontinuation.
5. Evidence of disease that may influence the outcome of the study within 4 weeks before dosing
6. Any history of abdominal surgery that may affect PK profiles of E2027
7. Any clinically abnormal symptom or organ impairment found by medical history, physical examinations, vital signs, ECG finding, or laboratory test results that requires medical treatment at Screening or Baseline
8. A prolonged QT/QTc interval (QTc greater than 450 ms) demonstrated on ECG at Screening or Baseline
9. Persistent systolic blood pressure greater than 130 mmHg or diastolic blood pressure greater than 85 mm Hg at Screening or Baseline (Parts A, B, and D)
10. Persistent systolic blood pressure greater than 140 mmHg or diastolic blood pressure greater than 90 mm Hg at Screening or Baseline (Part C)
11. Heart rate less than 50 or more than 100 beats/min at Screening or Baseline
12. History of prolonged QT/QTc interval
13. Left bundle branch block
14. History of myocardial infarction or active ischemic heart disease
15. History of clinically significant arrhythmia or uncontrolled arrhythmia
16. Known history of clinically significant drug allergy at Screening or Baseline
17. Known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening or Baseline
18. Known to be human immunodeficiency virus (HIV) positive at Screening
19. Active viral hepatitis (A, B or C) as demonstrated by positive serology at Screening
20. History of drug or alcohol dependency or abuse within the 2 years before Screening, or those who have a positive urine drug or alcohol test at Screening or Baseline
21. Intake of caffeinated beverages or food within 72 hours before dosing
22. Intake of nutritional supplements, juice, and herbal preparations or other foods or beverages that may affect the various drug metabolizing enzymes and transporters within 1 week before dosing
23. Intake of herbal preparations containing St. John's Wort within 4 weeks before dosing
24. Use of prescription drugs within 4 weeks before dosing
25. Intake of over-the-counter (OTC) medications within 2 weeks before dosing
26. Currently enrolled in another clinical trial or used any investigational drug or device within 30 days (or 5 half-lives, whichever is longer) preceding informed consent
27. Engagement in strenuous exercise within 2 weeks before check-in (eg, marathon runners, weight lifters, etc.)
28. Any contraindication to continuous CSF sampling via indwelling lumbar catheter (Part B only)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From screening up to 10 days
Plasma PK assessments of E2027 and its metabolites for Part A, Part B, Part C, and Part D - Cmax (maximum drug concentration) | Day 1 at predose and postdose 0.5 (30 minutes) to 18 hours, postdose on Day 2 (24 and 36 hours (parts A, B, C, D) and 30 hours (part B only), Day 3 (48 hours), Day 4 (72 hours), Day 5, (96 hours), Day 6 (120 hours), Day 7 (144 hours), Day 10 (216 hours)
  For participants in Part B of the 2nd cohort only, samples will also be collected on the following days of Treatment Period 2: Day 1 at predose and postdose 0.5 (30 minutes), 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 18 hours. Participants will receive a single oral dose of the same study drug that they received in the previous treatment period, but after a high-fat meal.
Plasma PK assessments of E2027 and its metabolites for Part A, Part B, Part C, and Part D - tmax (time to reach maximum (peak) concentration following drug administration) | Day 1 at predose and postdose 0.5 (30 minutes) to 18 hours, postdose on Day 2 (24 and 36 hours (parts A, B, C, D) and 30 hours (part B only), Day 3 (48 hours), Day 4 (72 hours), Day 5, (96 hours), Day 6 (120 hours), Day 7 (144 hours), Day 10 (216 hours)
  For participants in Part B of the 2nd cohort only, samples will also be collected on the following days of Treatment Period 2: Day 1 at predose and postdose 0.5 (30 minutes), 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 18 hours. Participants will receive a single oral dose of the same study drug that they received in the previous treatment period, but after a high-fat meal.
Plasma PK assessments of E2027 and its metabolites for Part A, Part B, Part C, and Part D - AUC (area under the concentration-time curve) | Day 1 at predose and postdose 0.5 (30 minutes) to 18 hours, postdose on Day 2 (24 and 36 hours (parts A, B, C, D) and 30 hours (part B only), Day 3 (48 hours), Day 4 (72 hours), Day 5, (96 hours), Day 6 (120 hours), Day 7 (144 hours), Day 10 (216 hours)
  For participants in Part B of the 2nd cohort only, samples will also be collected on the following days of Treatment Period 2: Day 1 at predose and postdose 0.5 (30 minutes), 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 18 hours. Participants will receive a single oral dose of the same study drug that they received in the previous treatment period, but after a high-fat meal.
Plasma PK assessments of E2027 and its metabolites for Part A, Part B, Part C, and Part D - t1/2 (terminal elimination half-life following last dose) | Day 1 at predose and postdose 0.5 (30 minutes) to 18 hours, postdose on Day 2 (24 and 36 hours (parts A, B, C, D) and 30 hours (part B only), Day 3 (48 hours), Day 4 (72 hours), Day 5, (96 hours), Day 6 (120 hours), Day 7 (144 hours), Day 10 (216 hours)
  For participants in Part B of the 2nd cohort only, samples will also be collected on the following days of Treatment Period 2: Day 1 at predose and postdose 0.5 (30 minutes), 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 18 hours. Participants will receive a single oral dose of the same study drug that they received in the previous treatment period, but after a high-fat meal.
Plasma PK assessments of E2027 and its metabolites for Part A, Part B, Part C, and Part D - CL/F (Apparent total clearance following extravascular (eg, oral) administration) | Day 1 at predose and postdose 0.5 (30 minutes) to 18 hours, postdose on Day 2 (24 and 36 hours (parts A, B, C, D) and 30 hours (part B only), Day 3 (48 hours), Day 4 (72 hours), Day 5, (96 hours), Day 6 (120 hours), Day 7 (144 hours), Day 10 (216 hours)
  Plasma PK assessments of E2027 and its metabolites for Part A, Part B and Part C - AUC Metabolite Ratio (Metabolite to E2027 ratio for AUC(0-inf) following molecular weight correction)
  For participants in Part B of the 2nd cohort only, samples will also be collected on the following days of Treatment Period 2: Day 1 at predose and postdose 0.5 (30 minutes), 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 18 hours. Participants will receive a single oral dose of the same study drug that they received in the previous treatment period, but after a high-fat meal.
Plasma PK assessments of E2027 and its metabolites for Part A, Part B, Part C, and Part D - Vz/F (Apparent volume of distribution at terminal phase) | Day 1 at predose and postdose 0.5 (30 minutes) to 18 hours, postdose on Day 2 (24 and 36 hours (parts A, B, C, D) and 30 hours (part B only), Day 3 (48 hours), Day 4 (72 hours), Day 5, (96 hours), Day 6 (120 hours), Day 7 (144 hours), Day 10 (216 hours)
  For participants in Part B of the 2nd cohort only, samples will also be collected on the following days of Treatment Period 2: Day 1 at predose and postdose 0.5 (30 minutes), 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 18 hours. Participants will receive a single oral dose of the same study drug that they received in the previous treatment period, but after a high-fat meal.
Plasma PK assessments of E2027 and its metabolites for Part A, Part B, Part C, and Part D - AUC Metabolite Ratio (Metabolite to E2027 ratio for AUC following molecular weight correction) | Day 1 at predose and postdose 0.5 (30 minutes) to 18 hours, postdose on Day 2 (24 and 36 hours (part A, B, C, D) and 30 hours (part B only), Day 3 (48 hours), Day 4 (72 hours), Day 5, (96 hours), Day 6 (120 hours), Day 7 (144 hours), Day 10 (216 hours)
  For participants in Part B of the 2nd cohort only, samples will also be collected on the following days of Treatment Period 2: Day 1 at predose and postdose 0.5 (30 minutes), 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 18 hours. Participants will receive a single oral dose of the same study drug that they received in the previous treatment period, but after a high-fat meal.
Urine PK assessments of E2027 and its metabolites for Part A and Part C - Ae (cumulative amount of drug excreted in urine up to 96 hours postdose) | Day 1 to Day 5 postdose at 0 to 4 hours and greater than 4 to 8 hours, 8 to 12 hours, 12 to 24 hours, 24 to 48 hours, 48 to 72 hours and 72 to 96 hours
Urine PK assessments of E2027 and its metabolites for Part A and Part C - CLR (renal clearance) | Day 1 to Day 5 postdose at 0 to 4 hours and greater than 4 to 8 hours, 8 to 12 hours, 12 to 24 hours, 24 to 48 hours, 48 to 72 hours and 72 to 96 hours
CSF PK assessments of E2027 and its metabolites for Part B - Cmax (maximum drug concentration) | At predose (0 hour), and postdose at 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 24 and 30 hours
CSF PK assessments of E2027 and its metabolites for Part B - tmax (time to reach maximum (peak) concentration following drug administration) | At predose (0 hour), and postdose at 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 24 and 30 hours
CSF PK assessments of E2027 and its metabolites for Part B - AUC (area under the concentration-time curve from zero time extrapolated to infinite time) | At predose (0 hour), and postdose at 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 24 and 30 hours
CSF PK assessments of E2027 and its metabolites for Part B - t1/2 (terminal elimination half-life following last dose) | At predose (0 hour), and postdose at 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 24 and 30 hours
CSF PK assessments of E2027 and its metabolites for Part B - CSF:plasma ratio (ratio of AUC for CSF:plasma) | At predose (0 hour), and postdose at 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 24 and 30 hours
PD assessments for Part B - change from baseline in CSF cGMP | At -3, - 2, -1 hours, predose (0 hour), and postdose at 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 24 and 30 hours
PD assessments for Part B - Amax (maximum change (%) of CSF cGMP concentration compared to baseline at a single time point within 30 hours postdose) | At -3, - 2, -1 hours, predose (0 hour), and postdose at 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 24 and 30 hours
PD assessments for Part B - tAmax (time at which Amax occurs for CSF cGMP) | At -3, - 2, -1 hours, predose (0 hour), and postdose at 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 24 and 30 hours
PD assessments for Part B - AUAC(-3 - 0 h) (area under the CSF cGMP concentration x time curve from time - 3 h to 0 h) | At -3, - 2, -1 hours, predose (0 hour), and postdose at 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 24 and 30 hours
PD assessments for Part B - AUAC(0 -30 h) (Area under the CSF cGMP concentration x time curve from time 0 h to 30 h) | At -3, - 2, -1 hours, predose (0 hour), and postdose at 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 24 and 30 hours
PD assessments for Part B -Delta AUAC(0 - 30 h) (Change (%) in AUAC averaged over 30 hours postdose relative to baseline AUAC averaged over 3 h predose for CSF cGMP, i.e. (AUAC(0 - 30 h)/30 minus AUAC(-3 - 0 h)/3)/(AUAC(-3 - 0 h)/3) | At -3, - 2, -1 hours, predose (0 hour), and postdose at 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 24 and 30 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Paraxel International, Glendale, California, United States